CLINICAL TRIAL: NCT01665092
Title: Phase 2 Study of Levo-Carnitine for Vasopressor Dependent Septic Shock
Brief Title: Rapid Administration of Carnitine in sEpsis
Acronym: RACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Alan Jones, Professor of Emergency Medicine, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GM103799
Record Dates: First submitted 2012-08-11; First posted 2012-08-15 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (Placebo Comparator): Normal saline
  Interventions: Drug: placebo
- Carnitine Low (Experimental): Levo-Carnitine 6g
  Interventions: Drug: Levo-Carnitine
- Carnitine Medium (Experimental): Levo-Carnitine 12 g
  Interventions: Drug: Levo-Carnitine
- Carnitine High (Experimental): Levo-Carnitine 18 g
  Interventions: Drug: Levo-Carnitine

INTERVENTIONS:
Drug: Levo-Carnitine
  Arms: Carnitine High; Carnitine Low; Carnitine Medium
Drug: placebo
  Arms: Control

SUMMARY:
Prior work has shown that exogenous L-carnitine administration enhances glucose and lactate oxidation, attenuates fatty acid toxicity, and improves endothelial-smooth muscle coupling and cardiac mechanical efficiency. The overall goal of this proposal is to investigate L-carnitine as a novel adjunctive treatment of septic shock. In this study the investigators will test our primary hypothesis: Early adjunctive L-carnitine administration in vasopressor dependent septic shock will significantly reduce cumulative organ failure at 48 hours with an associated decrease in 28-day mortality suggesting the need for further phase III study. To accomplish this the investigators will conduct a phase II, double blinded, placebo controlled, adaptive randomized trial of 250 eligible patients with vasopressor-dependent septic shock. Study subjects will be assigned to one of four arms: low (6g), medium (12g) or high (18g) dose intravenous L-carnitine or placebo for 12 hours as a part of early resuscitative care.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected or confirmed infection (examples include but are not limited to: white cells in a normally sterile body fluid; perforated viscus; radiographic evidence of pneumonia in clinical symptoms; a syndrome associated with a high risk of infection e.g. cellulitis, cutaneous abscess, ascending cholangitis, toxic shock syndrome, fever of unknown origin with high suspicion of infectious etiology)
2. Any two of four criteria of systemic inflammatory response as defined by the 2001 ACCP/SCCM Consensus Conference Committee;
3. Recognition of septic shock and initiation of quantitative resuscitation within 24 hours of enrollment;
4. Requirement of high dose vasopressors for ≥4 hours to treat shock: Norepinephrine > 0.05mcg/kg/min; dopamine >10mcg/kg/min; Phenylephrine >0.4 mcg/kg/min; epinephrine > 0.05 mcg/kg/min;
5. Cumulative sequential organ failure assessment (SOFA) score of ≥ 6;
6. Blood lactate level of >2.0 mMol/L.

Exclusion Criteria:

1. Age <18 years;
2. Pregnancy or breastfeeding;
3. Any primary diagnosis other than sepsis;
4. Established Do Not Resuscitate status or advanced directives restricting aggressive care or treating physician deems aggressive care unsuitable;
5. Any history of seizures or a known seizure disorder;
6. Any known inborn error of metabolism;
7. Anticipated requirement for surgery that would interfere with the 12 hour infusion time;
8. Active participation in another interventional study;
9. Cardiopulmonary resuscitation (chest compression or defibrillation) prior to enrollment;
10. Known systemic allergy to L-carnitine.
11. Severe immunocompromised state (e.g. subject has neutropenia [receiving cytotoxic chemotherapy with absolute neutrophil count <500/uL or expected to decline to < 500 uL within the next three days).
12. Active Treatment with Coumadin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2013-01; Primary Completion 2018-03 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Jones, MD, Principal Investigator — University of Mississippi Medical Center
Locations (14):
- United States (14):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Univeristy of California Davis, Sacramento, California
  - Christiana Care Health Services, Wilmington, Delaware
  - University of Florida, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - BIDMC, Boston, Massachusetts
  - BWH, Boston, Massachusetts
  - MGH, Boston, Massachusetts
  - St. Vincent Hospital, Worcester, Massachusetts
  - Wayne State University, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cooper University Hospital, Camden, New Jersey
  - Carolinas Medical Center, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jones AE, Puskarich MA, Shapiro NI, Guirgis FW, Runyon M, Adams JY, Sherwin R, Arnold R, Roberts BW, Kurz MC, Wang HE, Kline JA, Courtney DM, Trzeciak S, Sterling SA, Nandi U, Patki D, Viele K. Effect of Levocarnitine vs Placebo as an Adjunctive Treatment for Septic Shock: The Rapid Administration of Carnitine in Sepsis (RACE) Randomized Clinical Trial. JAMA Netw Open. 2018 Dec 7;1(8):e186076. doi: 10.1001/jamanetworkopen.2018.6076. PMID 30646314

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Normal saline
  placebo
- Carnitine Low: Levo-Carnitine 6g
  Levo-Carnitine
- Carnitine Medium: Levo-Carnitine 12 g
  Levo-Carnitine
- Carnitine High: Levo-Carnitine 18 g
  Levo-Carnitine
Period: Overall Study
Arm/Group | Control | Carnitine Low | Carnitine Medium | Carnitine High
Started | 75 | 35 | 34 | 106
Completed | 75 | 35 | 32 | 105
Not Completed | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Carnitine Low | Carnitine Medium | Carnitine High | Total
Number analyzed (Participants) | 75 | 35 | 34 | 106 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.22 (16.5) | 67.51 (12.01) | 64.91 (12.56) | 59.67 (14.50) | 62 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 17 | 13 | 42 | 108
  Male | 39 | 18 | 21 | 64 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3 | 6 | 12
  Not Hispanic or Latino | 72 | 35 | 31 | 100 | 238
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 75 | 35 | 34 | 106 | 250

OUTCOME MEASURES:

1. Primary Outcome: Delta SOFA Score
Description: Sequential Organ Failure Assessment Score (0-24 range). Delta SOFA is calculated as (SOFA Score at 48 hours post enrollment minus SOFA Score at enrollment). A negative value indicates improvement in the score.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Carnitine Low | Carnitine Medium | Carnitine High
Number analyzed (Participants) | 75 | 35 | 34 | 106
units on a scale | -1.8 (0.35) | -0.34 (0.66) | -1.68 (0.61) | -2.15 (0.37)

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Control | Carnitine Low | Carnitine Medium | Carnitine High
All-Cause Mortality (participants affected / at risk) | 34/75 | 20/35 | 16/34 | 45/106
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/35 | 0/34 | 0/106
Other Adverse Events (participants affected / at risk) | 0/75 | 0/35 | 0/34 | 0/106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/92/NCT01665092/Prot_SAP_000.pdf